CLINICAL TRIAL: NCT06488300
Title: Assessment of Respiratory SYNcytial Virus antivirALs: A Phase 2 Multi-centre Adaptive Randomised Platform Trial For the Assessment of Antiviral Pharmacodynamics in aCute Symptomatic RSV Infection (ARSYNAL-FC)
Brief Title: Assessing Antiviral Treatments in Early Symptomatic RSV
Acronym: ARSYNAL-FC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR24001
Record Dates: First submitted 2024-06-19; First posted 2024-07-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus; Respiratory Syncytial Virus, Human
Keywords: Respiratory Syncytial Virus; Phase 2; Antiviral Pharmacodynamics
MeSH Terms: interventions — Ribavirin; molnupiravir; favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Negative control group (No Intervention): Controls will receive no antiviral treatment (supportive treatment will remain the same as per the treating Physician's judgement)
- Ribavirin (Experimental): [Pending addition]
  Interventions: Drug: Ribavirin
- Molnupiravir (Experimental)
  Interventions: Drug: Molnupiravir
- Favipiravir (Experimental): [Pending addition]
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Ribavirin — Oral ribavirin 400 to 1000mg three times a day for 5 days. Each tablet contains 200mg, The total daily dosage in adults is weight dependent as outlined below;
  * 40-59.9kg = 1200mg/day
  * 60-79.9kg = 1800mg/day
  * 80-99.9kg = 2400mg/day
  * ≥100kg = 3000mg/day
  Arms: Ribavirin
Drug: Molnupiravir — Oral molnupiravir 800mg BD for 5 days
  Arms: Molnupiravir
Drug: Favipiravir — Oral favipiravir 1800mg BD on Day 0, and 800mg BD for a further 4 days
  Arms: Favipiravir

SUMMARY:
This trial will use a previously validated platform, to quantitatively assess antiviral effects in low-risk patients with high viral burdens and uncomplicated Respiratory Syncytial Virus (RSV), to determine in-vivo antiviral activity. In this randomised, open-label, controlled, group sequential adaptive platform trial, we will assess and compare the performance of currently licensed interventions (including repurposed drugs) with activity against RSV, and those with potential activity demonstrated in pre-clinical and early clinical studies relative to each-other, and the control (no antiviral treatment).

ARSYNAL-FC study is funded by Wellcome Trust Grant ref: 226933/Z/23/Z through the COVID-19 Therapeutics Accelerator

DETAILED DESCRIPTION:
There are no proven effective drug treatments for RSV. While vaccines are becoming available, and monoclonal antibodies exist for prevention in infants, antiviral treatments are still urgently needed.

The study is a randomised, open label, controlled, adaptive platform trial that will be conducted in low-risk adult patients (18 - <65 years old) with early symptomatic RSV, recruited from outpatient acute respiratory infection clinics (ARIs), other approved facilities, or by patient self-referral to the study site. The primary pharmacodynamic measure in this study is the rate of viral clearance following treatment. Individual patient's involvement for this study is 28 days.

This platform will compare antivirals with potential RSV antiviral activity, against a negative control (no treatment). Currently, interventions included in the platform are;

* Interventions licensed for paediatric RSV infections: ribavirin.
* Interventions with antiviral activity against RSV demonstrated in in-vitro studies: molnupiravir and favipiravir

Randomisation to the no antiviral treatment control arm (no intervention) will be fixed at a minimum of 20% throughout the study. The randomisation ratios will be uniform for all available interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient understands the procedures and requirements and is willing and able to give informed consent for full participation in the study
* Adults, male or female, aged ≥18 to <65 years at time of consent
* Early symptomatic RSV; at least one reported symptom of RSV (including fever, history of fever, myalgias, headache, cough, fatigue, nasal congestion, rhinorrhoea and sore throat) within 4 days (96 hours)
* RSV positive by rapid antigen test OR a positive RT-PCR test for RSV viruses within the last 24hrs with a Ct value of <30
* Able to walk unaided and unimpeded in activities of daily living (ADLs)
* Agrees and is able to adhere to all study procedures, including availability and contact information for follow-up visits

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

* Taking any concomitant medications or drugs which could interact with the study medications or have antiviral activity
* Presence of any chronic illness/condition requiring long term treatment or other significant comorbidity
* BMI ≥35 Kg/m2
* Clinically relevant laboratory abnormalities discovered at screening

  * Haemoglobin <10g/dL (<12g/dL for all arms if Ribavirin is in the randomisation)
  * Platelet count <100,000/uL
  * ALT > 2x ULN
  * Total bilirubin >1.5 x ULN
  * eGFR <70mls/min/1.73m2
* For females: pregnancy, actively trying to become pregnant or lactating (women on OCP are eligible to join)
* Contraindication to taking, or known hypersensitivity reaction to any of the proposed therapeutics
* Currently participating in another interventional RSV, influenza or COVID-19 therapeutic trial
* Clinical evidence of pneumonia- e.g., shortness of breath, hypoxaemia, crepitations (imaging not required)
* Known to be currently co-infected with influenza or SARS-CoV-2 (i.e. confirmed with positive ATK or RT-PCR)
* Received any RSV vaccine within the last year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of viral clearance for interventions relative to no study drug arm (superiority comparison) | Days 0-5
  Rate of viral clearance- estimated from the log10 viral density derived from qPCR of standardised duplicate oropharyngeal swabs taken daily from baseline (day 0) to day 5 for each therapeutic arm compared with the contemporaneous no antiviral treatment control/ positive control

SECONDARY OUTCOMES:
Rate of RSV clearance in early infection | Days 0-5
  Rate of viral clearance in early RSV infection to characterise the determinants of RSV clearance in early infection e.g., contribution of baseline serology, virus type/subtype, prior vaccination, host genetics
Rate of RSV clearance for drugs with evidence of antiviral activity | Days 0-5
  Rate of viral clearance to determine optimal dosing regimens for drugs with evidence of antiviral activity
Assessment of time to symptom alleviation across interventions | Days 0-14
  Time to symptom resolution across interventions
Assessment of fever duration across interventions | Days 0-14
  Area under the curve of recorded temperature across interventions
Effects of drugs on the development of drug resistant viral mutants | Days 0-14
  To determine the effects of drugs on the development of drug resistant viral mutants between intervention and no treatment arm, measuring the number of mutations known to confer resistance in detectable virus at later time points

OTHER OUTCOMES:
Hospitalisation for clinical reasons | Days 0-28
  To characterise the relationship between viral clearance and hospitalisation for clinical reasons up to day 28
Number of participants with virus-related complications | Days 0-28
  Number of participants with virus-related complications including bronchitis, sinusitis, otitis media and pneumonia requiring antibiotics, up to day 28, where the diagnosis is made and documented by the study clinician.

CONTACTS AND LOCATIONS:
Locations (2):
- Laos-Oxford-Mahosot Hospital-Wellcome Trust Research Unit, Vientiane, Laos
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With patient's consent, clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future. https://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies).
Access Criteria: Refer to MORU data sharing policy with other researchers to use in the future. https://wellcome.ac.uk/press-release/statement-data-sharing-public-health-emergencies).
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs